CLINICAL TRIAL: NCT03472534
Title: A 21-Day, Randomized, Controlled Study to Evaluate the Skin Irritation Potential of CCP-020 (Diacerein 1%) Topical Ointment in Healthy Subjects Using a Cumulative Irritant Patch Test Design
Brief Title: A 21 Day Irritation Study in Healthy Volunteers With Diacerein 1% Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Castle Creek Pharmaceuticals, LLC (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCP-020-102
Record Dates: First submitted 2018-01-30; First posted 2018-03-21 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — diacerein; Ointments

STUDY DESIGN:
Intervention Model Description: Cumulative irritancy patch test (CIPT) procedure. All subjects received once daily applications of 0.2mL of diacerein 1% ointment under occlusive patch for 21 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- study in healthy volunteers (Other): diacerein 1% ointment
  Interventions: Drug: diacerein 1% ointment

INTERVENTIONS:
Drug: diacerein 1% ointment — diacerein 1% ointment applied to the skin of the infrascapular area of the back under occlusive patch for 21 days.
  Other Names: CCP-020

SUMMARY:
Single center, randomized, controlled, evaluator blinded, within-subject study to evaluate the irritation potential of diacerein1% ointment on normal skin of healthy volunteers, using a cumulative irritancy patch test (CIPT) procedure.

DETAILED DESCRIPTION:
This study was designed to assess the cumulative irritation potential of diacerein 1% ointment in comparison with vehicle ointment, 0.2% sodium lauryl sulfate (SLS) (positive control), and 0.9% saline (negative control) on normal skin of healthy volunteers using a cumulative irritancy patch test (CIPT) procedure applied once daily for 21 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Is a healthy male or female (to be confirmed by medical history);
* Is 18 years of age or older;
* In the case of a female of childbearing potential, is using two acceptable forms of birth control;
* In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) on Day 1 prior to randomization and are willing to submit to a UPT at the end of study (EOS);
* Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs;
* Is of any Fitzpatrick Skin Type or race, providing the skin pigmentation will allow discernment of erythema

Key Exclusion Criteria:

* Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction;
* Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
* Is not willing to refrain from using systemic/topical anti-inflammatory analgesics such as aspirin, (occasional use of acetaminophen will be permitted);
* Is using medication which, in the opinion of the Investigator, will interfere with the study results;
* Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study;
* Has psoriasis and/or active atopic dermatitis/eczema;
* Has a known sensitivity or allergy to constituents of the materials being evaluated including diacerein, mineral oil, petrolatum, cetyl alcohol, D&C Yellow #10 and/or ethyl paraben;
* Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
* Has received treatment for any type of internal cancer within 5 years prior to study entry;
* Has any known sensitivity to adhesives; and/or
* Has received any investigational drug(s) within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Chair — Castle Creek Pharmaceuticals, LLC
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This does not apply
Units Other Than Participants: skin patch test sites
Groups:
- Single Cohort (Healthy Volunteers): Diacerein 1% ointment, vehicle ointment, 0.2% sodium lauryl sulfate (SLS; positive control), and 0.9% saline (negative control) were applied at 4 randomly assigned, adjacent skin sites on the infrascapular area of each subject's back once daily for 21 consecutive days.
Period: Overall Study
Arm/Group | Single Cohort (Healthy Volunteers)
Started | 46; 184 skin patch test sites (Each participant receives all 4 unit interventions.)
Diacerein 1% Ointment | 46; 46 skin patch test sites
Vehicle Ointment | 46; 46 skin patch test sites
0.2% Sodium Lauryl Sulfate (SLS) | 46; 46 skin patch test sites
0.9% Saline | 46; 46 skin patch test sites
Completed | 35; 140 skin patch test sites
Not Completed | 11; 44 skin patch test sites
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Cohort (Healthy Volunteers)
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Count of Participants: American Indian or Alaska Native | 0
  Count of Participants: Asian | 1
  Count of Participants: Native Hawaiian or Other Pacific Islander | 0
  Count of Participants: Black or African American | 27
  Count of Participants: White | 18
  Count of Participants: More than one race | 0
  Count of Participants: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Skin Irritation Score
Description: Evaluation of the sum of all subjects' cumulative irritation scores for 21 days at each patch site.
  Cumulative Irritation Score is a visual score rating the degree of erythema, edema, and other signs of cutaneous irritation: Minimum = 0; Maximum = 6; higher score is worse outcome.
Time Frame: Daily for 21 days
Population: Per Protocol Population includes all subjects who completed the study with 21 evaluations of irritancy or who discontinued patch sites due to limiting irritation, and was used for analysis of cumulative irritation.
Measure: Number; unit: Normalized cumulative irritation score
Units Other Than Participants: Patch sites
Arm/Group | Single Cohort (Healthy Volunteers)
Number analyzed (Participants) | 35
Number analyzed (Patch sites) | 140
Normalized cumulative irritation score
  Diacerein 1% ointment: number analyzed (Patch sites) | 35
  Diacerein 1% ointment | 0
  Vehicle 1% ointment: number analyzed (Patch sites) | 35
  Vehicle 1% ointment | 0
  0.2% sodium lauryl sulfate (SLS) (positive control: number analyzed (Patch sites) | 35
  0.2% sodium lauryl sulfate (SLS) (positive control | 339
  0.9% saline (negative control)" Arms/Groups): number analyzed (Patch sites) | 35
  0.9% saline (negative control)" Arms/Groups) | 15
Statistical Analysis 1: Comparison: Single Cohort (Healthy Volunteers); Test type: Other — The p-value for the overall F-test was used to determine if the mean irritation scores were equal for all four products; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event collection occurred from timing of first dose until completion of last study visit, i.e., 21 days.
Description: Adverse events were not assessed at a patch site-specific level.
Arm/Group | Single Cohort (Healthy Volunteers)
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

LIMITATIONS AND CAVEATS:
There were no limitations or caveats on this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT03472534/Prot_SAP_000.pdf